CLINICAL TRIAL: NCT03169244
Title: Efficacy and Safety of the Melanocortin Activator Bupropion in Treating Binge Drinking
Brief Title: Buproprion for Binge Drinking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, James Garbutt, MD, Professor of Medicine, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-1064; 1R21AA025186-01 (NIH)
Record Dates: First submitted 2017-05-11; First posted 2017-05-30 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Abuse
MeSH Terms: conditions — Alcoholism | interventions — Bupropion; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The design is a 1:1 random assignment to placebo or bupropion XL (300mg/d).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupropion (Active Comparator): Bupropion extended release
  Interventions: Drug: Bupropion
- Placebo (Placebo Comparator): Placebo oral tablet
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Bupropion — Bupropion XL will be initiated at 150 mg/d on Days 1-4 and increased to 300 mg/d for Days 5-84.
  Other Names: Wellbutrin Extended Release
  Arms: Bupropion
Drug: Placebo Oral Tablet — Placebo will be initiated on Day 1 and continue throughout the course of the study.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The present proposal is an innovative and translational clinical trial derived from exciting preclinical findings to test the hypothesis that treatment with the melanocortin activator bupropion can reduce binge drinking in humans. Furthermore, pilot data on moderating effects of coexisting nicotine use on the efficacy of bupropion for binge drinking population will be obtained. Evidence for an efficacy signal with good tolerability with this FDA approved medication would form the foundation to conduct a well-powered Phase II b trial. The development of an effective pharmacotherapy for binge drinking would be a significant clinical advance.

.

DETAILED DESCRIPTION:
The design is a 1:1 random assignment to placebo or bupropion XL (extended release) (300mg/d). The study biostatistician, will prepare the randomization schedule and include blocking by gender and nicotine dependence. Randomization will be based on a stratified block design, with gender and nicotine dependence as the stratification variables with medication/placebo randomly assigned in blocks of four.

Bupropion XL will be initiated at 150 mg/d on Days 1-4 and increased to 300 mg/d for Days 5-84. The University of North Carolina (UNC) Hospital's Investigational Drug Services (IDS) will prepare opaque capsules containing bupropion XL 150/300 mg and matching placebo. Capsules will be inserted into blister packs with each pack containing 1 week of medication. The IDS will receive the randomization schedule from our statistician and prepare the blister packs according to the blocked schedule with blocking for gender/nicotine dependence.

Recruitment, Telephone Screen, and Full Eligibility Screening: Subjects will initially be prescreened by phone and then at full screening read and sign the informed consent. A breathalyzer test will be administered (must be 0.00 gms/dl to give informed consent), height, weight and BMI recorded and a medical history and examination completed. Over-the-counter and prescription medication use will be recorded and nicotine use documented. Complete Blood Count (CBC) with differential; serum bilirubin, Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Gamma-Glutamyl Transferase (GGT,) sodium, potassium, chloride, blood urea nitrogen, creatinine, glucose; and urinalysis and urine toxicology completed. Women will be given a urine pregnancy test (Ub-HCG) at screening and at weeks 4, 8, and 12. Trained interviewers will conduct the psychiatric screening interview using the M.I.N.I. . The Structured Clinical Interview (SCID) Substance Use Disorders Module to establish Diagnostic and Statistical Manual (DSM-V) criteria for alcohol use disorders will be administered by one of the study doctors. The study coordinator will conduct the pretreatment 90-day Timeline Followback (TLFB) interview to identify amount of alcohol consumed and timeframe of consumption. A binge drinking episode requires a minimum of 5/4 (men/women) standard drinks consumed over about a two hour period, i.e. consuming a bottle of wine over five hours would not be coded as a binge drinking day. The Penn Alcohol Craving Scale (PACS) and the University of Rhode Island Change Assessment (URICA) will be completed and treatment goal-abstinence vs. reduction- recorded.

Initial Treatment Visit (within 21 days screening): Eligible individuals will not be required to abstain from drinking alcohol prior to randomization. The study coordinator will administer a breathalyzer test (BAC must be ≤0.04 gms/d) and complete assessments as outlined in Table 1, Protection of Human Subjects. A salivary cotinine sample will be taken A 1-week blister pack of bupropion-XL or placebo with written instructions will be dispensed from the Investigational Drug Services according to the randomization block along with a 1-week back-up blister pack in case of delayed appointments or lost doses. Bupropion-XL will be titrated with 150 mg given daily for 4 days followed by 300 mg/d. Participants will be given a calendar style diary to track pill taking, drinking quantity/timing, intoxication and any side effects. Finally, participants will receive Medical Management from a trained clinician.

Subsequent Treatment Visits: TLFB and PACS are gathered each visit, cotinine samples at weeks 4, 8 and 12 and URICA at week 8. Medical monitoring will be conducted by study physicians and will consist of review of vital signs, concomitant medication use, and general inquiries into side effects. The physician may recommend that medication be held for a period of time to deal with an adverse event, e.g. nausea. One month and three months following the last visit subjects will be contacted by phone to update drinking (TLFB), adverse effects and medications.

Medical Management Intervention: The psychosocial support for the study will be Medical Management (MM). MM sessions average 10-15 minutes and focus on three main areas: (1) feedback on consequences of drinking; (2) encouraging compliance with medication/addressing compliance problems and (3) encouraging progress towards drinking goal- reduction or abstinence are acceptable. 10% of sessions will be audiotaped and reviewed to enhance fidelity.

Medication Compliance Monitoring: Participants will record their pill taking in calendar-style diaries that will be provided and collected at each visit. Pills will be distributed in blister packs that will be returned to the study coordinator to reconcile any unused medication from the returned blister packs with participants' diary records.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 21 and 44 years.
2. A minimum of 5/3 (men/women) or more binge drinking episodes per month over the past three months. A binge drinking episode is defined as the consumption of 5/4 (men/women) standard drinks (~12 gms ethanol) in about a two hour period. Subjects may meet DSM-V criteria for mild or moderate alcohol use disorder.
3. Ability to understand and sign written informed consent.
4. Must have a 0.0 gms/dl breathalyzer reading on the day of screening and 0.0 gms/dl on the day of randomization.
5. BMI ≥18.5 (normal weight or above)
6. Express a desire to achieve abstinence or to reduce alcohol consumption
7. Must have a stable residence and be able to identify an individual who could contact participant if needed.

Exclusion Criteria:

1. Presence of physical dependence on alcohol as assessed by clear tolerance to alcohol or alcohol withdrawal symptoms based on SCID interview or a Severe Alcohol Use Disorder (>5 SCID DSM-V symptoms).
2. Bupropion is contraindicated in individuals with a history of bulimia or a seizure disorder
3. Clinically significant medical disease that might interfere with the evaluation of the study medication or present a safety concern (e.g., renal insufficiency, cirrhosis, unstable hypertension, diabetes mellitus, seizure disorder). Clinically significant psychiatric illness including any psychotic disorder, bipolar disorder, anorexia/bulimia, severe depression, or suicidal ideation.
4. Other substance abuse or dependence disorder other than nicotine or cannabis abuse.
5. Concurrent use of anticonvulsants. Concurrent use of any psychotropic medication including antidepressants, mood stabilizers, antipsychotics, anxiolytics, stimulants, or hypnotics with the exception of stable doses of antidepressants for one month. Bupropion is commonly added to antidepressants for augmentation so the use of another antidepressant does not represent a safety concern. .Prior history of adverse reaction to bupropion.
6. AST or ALT > 3.5 times Upper Limit of Normal (ULN) or bilirubin > 1.5 X ULN.
7. Positive urine toxicology screen with the exception of cannabis. Individuals with positive cannabis screens will be excluded only if they have a history of cannabis dependence.
8. Pregnant women and women of childbearing potential who do not practice a medically acceptable form of birth control (oral or depot contraceptive, or barrier methods such as diaphragm or condom with spermicidal).
9. Women who are breastfeeding.
10. Individuals requiring inpatient treatment or more intense outpatient treatment for their alcohol problems.
11. Participation in any clinical trial within the past 60 days that would have safety concerns for the trial.
12. Court-mandated participation in alcohol treatment or pending incarceration.

Ages: 21 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James C Garbutt, Principal Investigator — UNC Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupropion XL: Bupropion XL (extended release) will be initiated at 150 mg/d on Days 1-4 and increased to 300 mg/d for Days 5-84.
- Placebo: Placebo will be initiated on Day 1 and continue throughout the course of the study.
Period: Overall Study
Arm/Group | Bupropion XL | Placebo
Started | 22 | 20
Randomly Assigned | 22 | 20
Received Intervention | 22 | 18
Completed | 17 | 16
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupropion XL | Placebo | Total
Number analyzed (Participants) | 22 | 18 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.2 (7.26) | 24.4 (3.57) | 25.4 (5.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 19 | 15 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 18 | 40
Marital Status [Count of Participants; unit: Participants]
  Married | 3 | 3 | 6
  Divorced/Separated | 1 | 0 | 1
  Single, Never Married | 18 | 15 | 33
Years Education [Mean (Standard Deviation); unit: years] | 15.7 (2.27) | 16.2 (1.48) | 16.0 (1.95)
Smoking History [Count of Participants; unit: Participants] — Population: Data missing for two participants
  Participants
    Never Smoked: number analyzed (Participants) | 20 | 18 | 38
    Never Smoked | 17 | 15 | 32
    Less than or equal to 1/2 Pack/Day: number analyzed (Participants) | 20 | 18 | 38
    Less than or equal to 1/2 Pack/Day | 2 | 3 | 5
    Greater than or equal to 1 Pack/Day: number analyzed (Participants) | 20 | 18 | 38
    Greater than or equal to 1 Pack/Day | 1 | 0 | 1
Alcohol Use [Mean (Standard Deviation); unit: years] | 8.6 (6.02) | 7.2 (3.78) | 8.0 (5.12)
Mean Proportion Binge Drinking 90 Days Before Screening [Mean (Standard Deviation); unit: Proportion of Binge Drinking Days] — A Binge Drinking Day is defined as consumption of 5 (Male) or 4 (Female) standard alcohol drinks within a 2-hour period.
  Proportion of Binge Drinking Days | 0.27 (0.13) | 0.21 (0.09) | 0.24 (0.12)
Intensity per Binge Drinking Episode [Mean (Standard Deviation); unit: unitless] — Intensity is defined as the number of drinks per binge day scaled by the minimum threshold of a binge episode per gender (4 drinks/day for females; 5 drinks/day for males). Accordingly, if a female consumed 4 drinks in a binge drinking day, the intensity would be 1.0 and a female who consumed 6 drinks in a binge drinking day would have an intensity of 1.5.
  unitless | 1.64 (0.35) | 1.70 (0.53) | 1.67 (0.44)
Drinks per Binge Drinking Episode [Mean (Standard Deviation); unit: Drinks per Binge Episode] | 7.02 (1.31) | 7.24 (2.23) | 7.12 (1.76)
Gamma-glutamyltransferase (GGT) [Mean (Standard Deviation); unit: U/L] | 29.6 (23.8) | 25.0 (17.2) | 27.6 (21.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Proportion of Binge Drinking Days
Description: Frequency is assessed as number of binge episodes/time in trial controlling for missing data.
Time Frame: Randomization (Week 0) to Week 12
Population: Data unavailable for one placebo participant who did not provide any Timeline Follow Back data (TLFB).
Measure: Mean (Standard Deviation); unit: Binge Drinking Days
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 22 | 17
Binge Drinking Days | -0.13 (0.12) | -0.11 (0.09)

2. Primary Outcome: Change in the Intensity of Binge Drinking
Description: Intensity is defined as the number of drinks per binge day scaled by the minimum threshold of a binge episode per gender (4 drinks/day for females; 5 drinks/day for males). Accordingly, if a female consumed 4 drinks in a binge drinking day, the intensity would be 1.0 and a female who consumed 6 drinks in a binge drinking day would have an intensity of 1.5.
Time Frame: Randomization (Week 0) to Week 12
Population: Data unavailable for one placebo participant who did not provide any Timeline Follow Back data (TLFB).
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 22 | 17
unitless | -0.02 (0.48) | -0.09 (0.41)

3. Secondary Outcome: Change in GGT
Description: Change in serum Gamma-glutamyltransferase (GGT) levels
Time Frame: Randomization (Week 0) to Week 12
Population: Data unavailable for one placebo participant who did not provide GGT data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Bupropion XL | Placebo
Number analyzed (Participants) | 22 | 17
U/L | 12.8 (67.3) | -1.8 (9.75)

ADVERSE EVENTS:
Time Frame: From randomization through study follow-up, a total of approximately 16 weeks
Arm/Group | Bupropion XL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 11/22 | 13/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupropion XL (N=22) | Placebo (N=18)
Headache (Nervous system disorders) | 3 (4) | 8 (9)
Decreased Appetite (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (7)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (General disorders) | 4 (4) | 1 (1)
Dry Mouth (General disorders) | 3 (3) | 1 (1)
Sweating (General disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT03169244/Prot_SAP_000.pdf